CLINICAL TRIAL: NCT05567146
Title: The Effect of Tele-Nursing Gamification Technique on Nutritional Behavior and Physical Activity Level of Adolescents
Brief Title: The Effect of Tele-Nursing Gamification Technique
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aksaray University (Other)
Collaborators: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, sevim uğur, lecturer, Aksaray University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Aksaray Universıty
Record Dates: First submitted 2022-08-18; First posted 2022-10-05 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Adolescent
Keywords: Nutrition; Adolescent; Gamification; Tele-Nursing; Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: It is an experimental study with randomized pretest-posttest control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Adolescents going to high school, Gamification technique is applied to the Intervention group for seven weeks.
  Intervention:gamification technique with tele-nursing
  Interventions: Behavioral: Experimental group
- Control group (No Intervention): Adolescents going to high school

INTERVENTIONS:
Behavioral: Experimental group — It is planned to use the social media platform WhatsApp application to carry out the study. technique of gamification will have content in the form of points, ranking, penalties and rewards, which are the basic principles of gamification.
  Studies have shown that these contents are effective techniques to increase the interest, encouragement, motivation and purpose of the participants.
  Other Names: gamification technique with tele-nursing
  Arms: Experimental group

SUMMARY:
Adolescent health, safety and well-being cause it to be considered as an important and priority problem in terms of public health, as it affects many parts of the society. In this study, it was aimed to determine the effect of the gamification technique performed with tele-nursing on the nutritional behavior and physical activity level of adolescents.

DETAILED DESCRIPTION:
In recent years, with the advancement and widespread use of technology, the decrease in physical activity and the fact that the energy taken is more than the energy spent has brought the risks of many non-communicable diseases (such as obesity, cardiovascular diseases, certain types of cancer and diabetes).

It has been determined that one out of every four adults in the world does not meet the internationally recommended physical activity levels and more than 80% of the adolescent population is not physically active enough.

According to researches, there are unhealthy eating attitudes and behaviors in children and adolescents. Especially weight gain due to unhealthy diet makes individuals more susceptible to chronic diseases that increase the risk of disease and death. The most basic principle accepted for protection from these diseases and for a healthy life is to change the lifestyle and eating habits at an early age. In this context, schools that are in constant contact with students have been the most popular settings to promote healthy eating and adequate physical activity.

Considering our society's need for health services; In addition to the advantages of tele-nursing such as being accessible and cheap, providing long-term follow-up and counseling with ease of application, providing quick solutions in the detection of early-term symptoms, reducing emergency service applications, increasing patient satisfaction, and saving in cost-effectiveness and health expenditures, especially in our recent experience. It is seen that tele-nursing applications should be used in school health services, with the least number of people in contact with and providing cost-effective service in the upcoming pandemic processes. In addition, it is emphasized that the use of gamification techniques is more promising to increase telehealth-based physical activity interventions and to provide permanent behavior change.

Gamification is the use of game design elements such as scores and levels. It has been found that the applications made with the gamification technique motivate individuals to change their behaviors, increase participation and have a lasting effect on healthy behavior change.

With this study, it is thought that various applications that can be made within the scope of tele-nursing can provide continuity in the provision of school health services, as well as guide health personnel and school administrators in future health service planning in gaining permanent health behaviors. In addition, the importance of using digital approaches to optimize public health practices during the Covid-19 pandemic has been understood more and more and will contribute to the literature for various applications that can be made with tele-nursing in reducing and controlling health problems in possible pandemic situations.

Objective: In this study, to determine the effect of tele-nursing gamification technique on the nutritional behavior and physical activity level of adolescents.

Methodology: This is an experimental study with randomized pretest-posttest control group. The sample consisted of 80 students (40 in the experimental group, 40 in the control group) studying at Somuncubaba Anatolian High School, Uluırmak Vocational and Technical High School and Abdülhamit Han Science High School located in the city center of Aksaray. The gamification technique was applied via tele-nursing. Data were collected using Descriptive Characteristics Form, Adolescents Physical Activity Scale (AFAI), Step Count Tracking Chart, Water Drinking Tracking Chart, Beverage Consumption Form, Fruit and Vegetable Consumption Change Process Scale (MSTSS), Nutritional Behavior Scale, Health Status Perception Scale. Interviews were conducted using the form-filling technique. The gamification technique will be performed for a total of 7 weeks.

ELIGIBILITY:
Inclusion Criteria:

* To be studying in high schools determined by lot in Aksaray city center
* Volunteering to participate in research
* Signing the pediatric voluntary consent form
* Permission of the student to participate in the research by the parent
* Having a smartphone and an active WhatsApp account

Exclusion Criteria:

* Implementing a regular exercise program
* To apply any diet program (diabetic, vegan, vegetarian, alkaline, ketogenic diet etc.)
* Having a chronic illness
* Using regular medication

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
Descriptive Characteristics Information Form | week 0
  It consists of a total of 10 questions, including three open-ended and seven multiple-choice questions.
Physical Activity Scale for Adolescents | week 0
  On the scale, 5 points indicate the highest level of physical activity and 1 point indicates the lowest level of physical activity. While the minimum score to be obtained from the scale is 8, the highest score is 40. It is considered low when the physical activity level approaches 8 and high when it approaches 40.
Beverage Consumption Form | week 0
  daily drink types and quantities are recorded
Fruit and Vegetable Consumption Change Process Scale | week 0
  The scale is in a 5-point Likert type and each item is scored from 1 to 5. "Reflecting on the last month, indicate how much you agree with the following statements?" the question is; It is answered by marking one of the answer options such as 1"I do not agree at all", 2 "I do not agree", 3 "I am undecided", 4 "I partially agree", 5 "I completely agree". The highest score that can be obtained from the scale is 95, the lowest score is 19. Higher scores indicate a higher chance of succeeding in change.
Feeding Behavior Scale | week 0
  It measures children's heart health-promoting (low-fat and low-salt) food consumption habits. Children are shown comparable foods and asked which of the two foods they ate the most (frequently). A high total score from the scale indicates healthy eating habits. Scale items are -1 for unhealthy food and +1 for healthy food, the total score is between -14 and +14.
Health Status Perception Scale | week 0
  . The scale consists of a single item and the participants are asked to rate the question "How do you interpret your health at the moment". A score of 1 is given for the "very good" answer, 2 for the "good" answer, 3 for the "bad" answer, and 4 for the "very bad" answer. lowest score to be taken from the scale is 4 and the highest score is 1.

SECONDARY OUTCOMES:
Physical Activity Scale for Adolescents | 7 weeks
  On the scale, 5 points indicate the highest level of physical activity and 1 point indicates the lowest level of physical activity. While the minimum score to be obtained from the scale is 8, the highest score is 40. It is considered low when the physical activity level approaches 8 and high when it approaches 40.
Beverage Consumption Form | 7 weeks
  daily drink types and quantities are recorded
Fruit and Vegetable Consumption Change Process Scale | 7 weeks
  The scale is in a 5-point Likert type and each item is scored from 1 to 5. "Reflecting on the last month, indicate how much you agree with the following statements?" the question is; It is answered by marking one of the answer options such as 1"I do not agree at all", 2 "I do not agree", 3 "I am undecided", 4 "I partially agree", 5 "I completely agree". The highest score that can be obtained from the scale is 95, the lowest score is 19. Higher scores indicate a higher chance of succeeding in change.
Feeding Behavior Scale | 7 weeks
  It measures children's heart health-promoting (low-fat and low-salt) food consumption habits. Children are shown comparable foods and asked which of the two foods they ate the most (frequently). A high total score from the scale indicates healthy eating habits. Scale items are -1 for unhealthy food and +1 for healthy food, the total score is between -14 and +14.
Health Status Perception Scale | 7 weeks
  The scale consists of a single item and the participants are asked to rate the question "How do you interpret your health at the moment". A score of 1 is given for the "very good" answer, 2 for the "good" answer, 3 for the "bad" answer, and 4 for the "very bad" answer. lowest score to be taken from the scale is 4 and the highest score is 1.

CONTACTS AND LOCATIONS:
Overall Officials: sevim uğur, Principal Investigator — Aksaray University; özlem örsal, Study Director — Eskisehir Osmangazi University
Locations (1):
- Aksaray University, Aksaray, Centre, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No